CLINICAL TRIAL: NCT05301985
Title: Effects of Preoperative Oral Carbohydrate Loading on Neutrophil/Lymphocyte Ratio and Postoperative Complications Following Colorectal Cancer Surgery: a Randomized Controlled Study
Brief Title: Preoperative Administration of Oral Carbohydrate Drink, Neutrophil/Lymphocyte Ratio and Postoperative Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nermina Rizvanović (Other)
Responsible Party: Sponsor-Investigator, Nermina Rizvanović, PhD Anesthesiology and Intensive Care Specialist, Cantonal Hospital Zenica
Organization: Cantonal Hospital Zenica (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NR03/22
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Neutrophil; Lymphocyte; Postoperative Complications
Keywords: fasting; carbohydrate; colorectal carcinoma; nutritional status
MeSH Terms: conditions — Postoperative Complications; Fasting; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The patients with diagnosed colon cancer were hospitalized and prepared for elective, open colon surgery at the Department of Surgery. Before surgical procedure, the patients were undergoing to a preoperative anesthetic visit. During the visit, participants were assessed according to eligibility for enrollment in the study. The participants who have met the eligibility criteria have explained the nature of the study protocol. Those who agreed to participate in the study were randomized to one of two study groups for the duration of the study.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeons, anesthetists, and outcome assessors were masking to the treatment allocation.
  A nurse from the Department of Surgery performed the allocation into groups. The night before the operation, the nurse managed the patients according to the assigned intervention, but was not included in the study protocol. The next morning, the surgeon and anesthetist performed open elective colon surgery under general anesthesia, but without knowledge of the type of intervention.
  Independent outcomes assessors evaluated patients up to 30 days post-surgery and were also masked, without knowledge of the type intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting group (No Intervention): conventional preoperative fasting protocol The participants in the Fasting group stopped oral intake at 12:00 pm, the night before surgery. After surgery the participants fasted until the recovery of function of the bowel.
- Carbohydrate group (Experimental): preoperative nutrition The participants of experimental group consumed 400 ml of a clear carbohydrate drink (12,5 gr/100 ml carbohydrate, 50 kcal/100 ml, pH 5.0) at 10:00 pm the evening before surgery and 200 ml of the carbohydrate drink on the day of surgery, 2 hours before induction of anesthesia. After surgery the participants fasted until the recovery of function of the bowel.
  Interventions: Dietary Supplement: preoperative nutrition

INTERVENTIONS:
Dietary Supplement: preoperative nutrition — The participants of experimental group consumed 400 ml of a clear carbohydrate drink (12,5 gr/100 ml carbohydrate, 50 kcal/100 ml, pH 5.0) at 10:00 pm the evening before surgery and 200 ml of the carbohydrate drink on the day of surgery, 2 hours before induction of anesthesia. After surgery the participants fasted until the recovery of function of the bowel.
  Arms: Carbohydrate group

SUMMARY:
This study evaluated the impact of a preoperative carbohydrate oral drink on the postoperative Neutrophil / Lymphocyte Ratio (NLR) and the incidence of postoperative complications after elective open colon surgery compared to the conventional preoperative fasting protocol. Hypothesis was: preoperative carbohydrate loading reduces postoperative NLR value and reduces the incidence and severity of postoperative complications in colorectal surgery.

DETAILED DESCRIPTION:
This prospective randomized, controlled clinical study was carried out in the Department of Anesthesiology and Intensive Care Unit and Department of Surgery at the Cantonal Hospital Zenica, Bosnia and Herzegovina. The study protocol was approved by the local Ethics Committee.

A total of 60 participants who scheduled for elective open colon surgery and fulfilled study criteria were included into study. The purpose and procedures of the study were fully explained and voluntary, informed, written consent was obtained from each participant. The participants were randomly allocated into two equal groups, depending on the preoperative treatment. There were no reliable published data for effects of preoperative carbohydrate loading on postoperative NLR values. Based on our hypothesis, a pilot study was performed with ten patients per group. Mean postoperative NLR value was 8,67±4,98 in the participants with a conventional preoperative fasting protocol versus 4,76±2,83 in the participants with preoperative carbohydrate loading. Sample size was estimated using sample size calculator software and power analysis with 95% confidence interval and power of 80%. Statistical significance was considered as p< 0,05. The calculation indicated 27 participants per group would be sufficient to detect a difference of 3,91 with a standard deviation of 4,93 in NLR value between the groups. Assuming dropout of 10%, 30 participants per group were included. Block randomization was used with a block size of six and a 1:1 group ratio. A computer-generated random numbers indicating preoperative intervention, were sealed in opaque envelopes. An investigator who conducted randomization and opened the envelopes the night before surgery was blinded to the study protocol as well as the surgeons, nurses, anesthesiologists and staff involved in data collection.

The participants in the Fasting group (control group) stopped oral intake at 12:00 pm the night before surgery and underwent to a conventional preoperative fasting protocol. Participants in the Carbohydrate group (experimental group) consumed 400 ml of a clear carbohydrate solution at 10:00 pm the night before surgery and 200 ml of a clear carbohydrate solution, 2 hours prior induction of anesthesia. All participants underwent general anesthesia followed by colorectal surgery.

Fasting peripheral venous blood samples were collected at 06:00 am on the day of surgery (basal value), at 06:00 am on the first postoperative day, at 06:00 am on the third postoperative day and at 06:00 am on the fifth postoperative day. White blood counts were analysed with automated differential counts. The NLR value was obtained by dividing the absolute neutrophil count and the absolute lymphocyte count. All participants were followed up to 30 days post-surgery to assess postoperative complications and readmission rate. After discharge, participants were called by phone, once a week. Postoperative complications were graded for incidence and severity using the Clavien-Dindo Classification of Surgical Complications.

Demographic and surgical data of the participants were recorded: age, sex, body weight, body mass index, American Society of Anesthesiologists (ASA) physical status class, nutritional status of the participants according to Nutritional Risk Screening 2002 (NRS-2002), tumor localization and duration of surgery.

ELIGIBILITY:
Inclusion Criteria:

* participants with diagnosed colorectal carcinoma scheduled for elective open colorectal surgery
* aged between 18 years and 70 years
* participants with ASA physical status class I-III

Exclusion Criteria:

* previous treatment of colon, rectum or any other cancer
* emergency or palliative colon and rectum surgery
* disseminated malignant disease
* body mass index below 20 and above 30 kg/mᶺ2
* overall score ≥3 after final assessment of the nutritional status according to Nutritional Risk Screening 2002 (NRS-2002)
* disease with increased risk of aspiration
* history of diabetes mellitus
* history of hematological disease
* evidence of systemic inflammation
* immunomodulatory therapy
* neuromuscular disease
* pregnancy
* mental disease
* allergy to any study drugs
* alcoholic or drug abuse
* patient's refusal to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
The mean change in NLR values between conventional preoperative fasting protocol and a preoperative carbohydrate loading | fasting peripheral venous blood samples were collected at 06:00 am on the day of surgery (basal value), at 06:00 am on the first postoperative day, at 06:00 am on the third postoperative day and at 06:00 am on the fifth postoperative day.
  White blood counts with automated differential counts were analysed from peripheral venous blood samples using fluorescence flow cytometry method. The NLR value was calculated by following equation: NLR = the absolute neutrophil count (range of normality 4,0-7,0x10ᶺ9/L) / the absolute lymphocyte count (range of normality 1-3,7x10ᶺ9/L).
The mean change in delta NLR value between conventional preoperative fasting protocol and a preoperative carbohydrate loading | fasting peripheral venous blood samples were collected at 06:00 am on the day of surgery (basal value), at 06:00 am on the first postoperative day, at 06:00 am on the third postoperative day and at 06:00 am on the fifth postoperative day.
  Delta NLR value was defined as dynamic change in NLR value from basal value to the highest measured post-surgery NLR value. Delta NLR was calculated using following equation: Delta NRL = the highest measured post-surgery NLR value - basal NLR value.

SECONDARY OUTCOMES:
The mean change in incidence and severity of postoperative complications assessed using the Clavien-Dindo Classification of Surgical Complications between conventional preoperative fasting protocol and a preoperative carbohydrate loading | the incidence and severity of postoperative complications were assessed up to 30 days post-surgery. After discharge, participants were called by phone once a week and finally on the 30th day post-surgery.
  Postoperative complications were graded as follow: Grade I considered any deviation from the normal course without the need for pharmacological treatment or surgical, endoscopic and radiologic interventions. Grade II required pharmacological treatment with drugs other than such allowed for Grade I complications. Grade I and Grade II were considered minor postoperative complications. Grade III required surgical, endoscopic or radiological intervention without or with general anesthesia. Grade IV considered life-threatening complication required intensive care unit management. Grade V included death of patient. Grade III, IV and V were considered major complications.
The mean change in characteristics of postoperative complications between conventional preoperative fasting protocol and a preoperative carbohydrate loading | the characteristics of postoperative complications and readmission rate were assessed up to 30 days post-surgery. After discharge, participants were called by phone once a week and finally on the 30th day post-surgery.
  Characteristics of postoperative complications included: overall number of complications per group, number of participants without complications per group, number of participants with complications per group, number of participants with 1 complication per group, number of participants with 2 complications per group, number of participants with >2 complications per group and readmission rate per group within 30 days post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nermina Rizvanović, PhD, Principal Investigator — Cantonal Hospital Zenica, Crkvice 67, 72 000 Zenica, Bosnia and Herzegovina
Locations (1):
- Cantonal Hospital Zenica, Zenica, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Morrison CE, Ritchie-McLean S, Jha A, Mythen M. Two hours too long: time to review fasting guidelines for clear fluids. Br J Anaesth. 2020 Apr;124(4):363-366. doi: 10.1016/j.bja.2019.11.036. Epub 2020 Jan 17. No abstract available. PMID 31959387
- [Background] Vano YA, Oudard S, By MA, Tetu P, Thibault C, Aboudagga H, Scotte F, Elaidi R. Optimal cut-off for neutrophil-to-lymphocyte ratio: Fact or Fantasy? A prospective cohort study in metastatic cancer patients. PLoS One. 2018 Apr 6;13(4):e0195042. doi: 10.1371/journal.pone.0195042. eCollection 2018. PMID 29624591
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Sarin A, Chen LL, Wick EC. Enhanced recovery after surgery-Preoperative fasting and glucose loading-A review. J Surg Oncol. 2017 Oct;116(5):578-582. doi: 10.1002/jso.24810. Epub 2017 Aug 28. PMID 28846137
- [Background] Abola RE, Gan TJ. Preoperative Fasting Guidelines: Why Are We Not Following Them?: The Time to Act Is NOW. Anesth Analg. 2017 Apr;124(4):1041-1043. doi: 10.1213/ANE.0000000000001964. No abstract available. PMID 28319543
- [Background] Singh SM, Liverpool A, Romeiser JL, Miller JD, Thacker J, Gan TJ, Bennett-Guerrero E. A U.S. survey of pre-operative carbohydrate-containing beverage use in colorectal enhanced recovery after surgery (ERAS) programs. Perioper Med (Lond). 2021 May 28;10(1):19. doi: 10.1186/s13741-021-00187-3. PMID 34044894
- [Background] Ackerman RS, Tufts CW, DePinto DG, Chen J, Altshuler JR, Serdiuk A, Cohen JB, Patel SY. How Sweet Is This? A Review and Evaluation of Preoperative Carbohydrate Loading in the Enhanced Recovery After Surgery Model. Nutr Clin Pract. 2020 Apr;35(2):246-253. doi: 10.1002/ncp.10427. Epub 2019 Oct 21. PMID 31637778
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Background] Patel SY, Trona N, Alford B, Laborde JM, Kim Y, Li R, Manley BJ, Gilbert SM, Sexton WJ, Spiess PE, Poch MA. Preoperative immunonutrition and carbohydrate loading associated with improved bowel function after radical cystectomy. Nutr Clin Pract. 2022 Feb;37(1):176-182. doi: 10.1002/ncp.10661. Epub 2021 Apr 26. PMID 33900647
- [Background] Cheng PL, Loh EW, Chen JT, Tam KW. Effects of preoperative oral carbohydrate on postoperative discomfort in patients undergoing elective surgery: a meta-analysis of randomized controlled trials. Langenbecks Arch Surg. 2021 Jun;406(4):993-1005. doi: 10.1007/s00423-021-02110-2. Epub 2021 Feb 25. PMID 33629128
- [Background] Noba L, Wakefield A. Are carbohydrate drinks more effective than preoperative fasting: A systematic review of randomised controlled trials. J Clin Nurs. 2019 Sep;28(17-18):3096-3116. doi: 10.1111/jocn.14919. Epub 2019 Jun 10. PMID 31112338
- [Background] Liu X, Zhang P, Liu MX, Ma JL, Wei XC, Fan D. Preoperative carbohydrate loading and intraoperative goal-directed fluid therapy for elderly patients undergoing open gastrointestinal surgery: a prospective randomized controlled trial. BMC Anesthesiol. 2021 May 21;21(1):157. doi: 10.1186/s12871-021-01377-8. PMID 34020596
- [Background] Chen X, Li K, Yang K, Hu J, Yang J, Feng J, Hu Y, Zhang X. Effects of preoperative oral single-dose and double-dose carbohydrates on insulin resistance in patients undergoing gastrectomy:a prospective randomized controlled trial. Clin Nutr. 2021 Apr;40(4):1596-1603. doi: 10.1016/j.clnu.2021.03.002. Epub 2021 Mar 7. PMID 33752148
- [Background] Cook EJ, Walsh SR, Farooq N, Alberts JC, Justin TA, Keeling NJ. Post-operative neutrophil-lymphocyte ratio predicts complications following colorectal surgery. Int J Surg. 2007 Feb;5(1):27-30. doi: 10.1016/j.ijsu.2006.05.013. Epub 2006 Jun 27. PMID 17386911
- [Background] Mik M, Dziki L, Berut M, Trzcinski R, Dziki A. Neutrophil to Lymphocyte Ratio and C-Reactive Protein as Two Predictive Tools of Anastomotic Leak in Colorectal Cancer Open Surgery. Dig Surg. 2018;35(1):77-84. doi: 10.1159/000456081. Epub 2017 Jan 28. PMID 28132052
- [Background] Walker PA, Kunjuraman B, Bartolo DCC. Neutrophil-to-lymphocyte ratio predicts anastomotic dehiscence. ANZ J Surg. 2018 Jan 27. doi: 10.1111/ans.14369. Online ahead of print. PMID 29377500
- [Background] Mahsuni Sevinc M, Riza Gunduz U, Kinaci E, Armagan Aydin A, Bayrak S, Umar Gursu R, Gunduz S. Preoperative neutrophil-to-lymphocyte ratio and plateletto- lymphocyte ratio as new prognostic factors for patients with colorectal cancer. J BUON. 2016 Sept-Oct;21(5):1153-1157. PMID 27837617
- [Background] Li Z, Zhao R, Cui Y, Zhou Y, Wu X. The dynamic change of neutrophil to lymphocyte ratio can predict clinical outcome in stage I-III colon cancer. Sci Rep. 2018 Jun 21;8(1):9453. doi: 10.1038/s41598-018-27896-y. PMID 29930287
- [Background] Paliogiannis P, Deidda S, Maslyankov S, Paycheva T, Farag A, Mashhour A, Misiakos E, Papakonstantinou D, Mik M, Losinska J, Scognamillo F, Sanna F, Feo CF, Cherchi G, Xidas A, Zinellu A, Restivo A, Zorcolo L. Blood cell count indexes as predictors of anastomotic leakage in elective colorectal surgery: a multicenter study on 1432 patients. World J Surg Oncol. 2020 May 6;18(1):89. doi: 10.1186/s12957-020-01856-1. PMID 32375770
- [Background] Zhang YY, Li WQ, Li ZF, Guo XH, Zhou SK, Lin A, Yan WH. Higher Levels of Pre-operative Peripheral Lymphocyte Count Is a Favorable Prognostic Factor for Patients With Stage I and II Rectal Cancer. Front Oncol. 2019 Sep 24;9:960. doi: 10.3389/fonc.2019.00960. eCollection 2019. PMID 31612109
- [Background] Jakubowska K, Koda M, Kisielewski W, Kanczuga-Koda L, Grudzinska M, Famulski W. Pre- and postoperative neutrophil and lymphocyte count and neutrophil-to-lymphocyte ratio in patients with colorectal cancer. Mol Clin Oncol. 2020 Nov;13(5):56. doi: 10.3892/mco.2020.2126. Epub 2020 Aug 25. PMID 32905328
- [Background] Xia LJ, Li W, Zhai JC, Yan CW, Chen JB, Yang H. Significance of neutrophil-to-lymphocyte ratio, platelet-to-lymphocyte ratio, lymphocyte-to-monocyte ratio and prognostic nutritional index for predicting clinical outcomes in T1-2 rectal cancer. BMC Cancer. 2020 Mar 12;20(1):208. doi: 10.1186/s12885-020-6698-6. PMID 32164623
- [Background] Forget P, Dinant V, De Kock M. Is the Neutrophil-to-Lymphocyte Ratio more correlated than C-reactive protein with postoperative complications after major abdominal surgery? PeerJ. 2015 Jan 13;3:e713. doi: 10.7717/peerj.713. eCollection 2015. PMID 25653901
- [Background] Ozgehan G, Kahramanca S, Kaya IO, Bilgen K, Bostanci H, Guzel H, Kucukpinar T, Kargici H. Neutrophil-lymphocyte ratio as a predictive factor for tumor staging in colorectal cancer. Turk J Med Sci. 2014;44(3):365-8. doi: 10.3906/sag-1305-33. PMID 25558634
- [Background] Lobo DN, Gianotti L, Adiamah A, Barazzoni R, Deutz NEP, Dhatariya K, Greenhaff PL, Hiesmayr M, Hjort Jakobsen D, Klek S, Krznaric Z, Ljungqvist O, McMillan DC, Rollins KE, Panisic Sekeljic M, Skipworth RJE, Stanga Z, Stockley A, Stockley R, Weimann A. Perioperative nutrition: Recommendations from the ESPEN expert group. Clin Nutr. 2020 Nov;39(11):3211-3227. doi: 10.1016/j.clnu.2020.03.038. Epub 2020 Apr 18. PMID 32362485